CLINICAL TRIAL: NCT05923775
Title: Comparative Effectiveness of Preemptive Ibuprofen, Ketamine, and Their Combination in Postoperative Pain and Trismus Management Following Third Molar Surgery
Brief Title: Pain and Trismus Control in Third Molar Surgery: Ibuprofen, Ketamine, and Their Combination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cihan Topan (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Sponsor-Investigator, Cihan Topan, Assistant professor, Principal Investigator, Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/197
Record Dates: First submitted 2023-06-16; First posted 2023-06-28 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Molar, Third
Keywords: pain; trismus; analgesia; ketamine; Ibuprofen
MeSH Terms: conditions — Pain; Trismus; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intrafen group (Active Comparator): Each patient in this group will be administered intravenous Ibuprofen (400 mg/8 ml i.v. infusion) for pre-emptive analgesic effect 60 minutes before surgical third molar extraction. Before the procedure, each patient in this group will be given 2 ml of local anesthesia.
  Interventions: Procedure: Impacted third molar surgey
- Ketamine group (Active Comparator): Each patient in this group will be administered intravenous 100 ml saline (Poliflex 0.9% isotonic 100 ml solution) for a placebo effect 60 minutes before surgical third molar extraction. Before the procedure, each patient in this group will be given 0.3 mg/kg of ketamine (Ketalar 500 mg) in addition to 2 ml of local anesthesia.
  Interventions: Procedure: Impacted third molar surgey
- Combined group (Intrafen+Ketamine) (Active Comparator): Each patient in this group will be administered intravenous Ibuprofen (400 mg/8 ml i.v. infusion) for pre-emptive analgesic effect 60 minutes before surgical third molar extraction. Before the surgery, each patient in this group will be given 0.3 mg/kg of ketamine (Ketalar 500 mg) in addition to 2 ml of local anesthesia.
  Interventions: Procedure: Impacted third molar surgey
- Control (Placebo Comparator): Each patient in this group will be administered intravenous 100 ml saline (Poliflex 0.9% isotonic 100 ml solution) for a placebo effect 60 minutes before surgical third molar extraction. Before the procedure, each patient in this group will be given 2 ml of local anesthesia.
  Interventions: Procedure: Impacted third molar surgey

INTERVENTIONS:
Procedure: Impacted third molar surgey — The surgery was performed using the classic technique: ten minutes after anesthesia administration, a horizontal and sulcular incision was performed, and a mucoperiosteal envelope flap was elevated. The bone covering the impacted third molar tooth was removed with the use of a surgical handpiece and rotary instrument. During the operation, saline water was applied to the surgical drill with a second hand to protect the bone from developing a high temperature. After extraction of the third molar, the cavity was treated with curettage, irrigated with saline, and sutured.

SUMMARY:
The goal of the clinical trial is to compare the efficacy of ibuprofen, ketamine, and their combination in managing postoperative pain and trismus following third molar surgery. The main question it aims to answer is: which is the best way to control pain and trismus after third molar surgery?

DETAILED DESCRIPTION:
Materials and methods The study will comprise 100 individuals who requested to have their mandibular third molar tooth extracted at the Erciyes University Faculty of Dentistry. Participants were randomly allocated into four groups, with 25 patients in each group.

The first group (Intrafen group): Each patient in this group will be administered intravenous Ibuprofen (400 mg/8 ml i.v. infusion) for pre-emptive analgesic effect 60 minutes before surgical third molar extraction. Before the procedure, patients will be given local anesthesia using a mixture of 2 ml of local anesthetic (Ultracain Ds Fort 2 ml) plus 3 ml of saline solution (Poliflex 0.9% isotonic 100 ml solution). The impacted third molars of the patients will be removed.

The second group (Ketamine group): Each patient in this group will be administered intravenous 100 ml saline (Poliflex 0.9% isotonic 100 ml solution) for a placebo effect 60 minutes before surgical third molar extraction. Before the procedure, patients will be given local anesthesia using a mixture of 2 ml of local anesthetic (Ultracain Ds Fort 2 ml) plus 3 ml of saline solution (Poliflex 0.9% isotonic 100 ml solution) plus 0,3 mg/kg of ketamine (Ketalar 500 mg). The impacted third molars of the patients will be removed.

The third group (Combined group): Each patient in this group will be administered intravenous Ibuprofen (400 mg/8 ml i.v. infusion) for pre-emptive analgesic effect 60 minutes before surgical third molar extraction. Before the procedure, patients will be given local anesthesia using a mixture of 2 ml of local anesthetic (Ultracain Ds Fort 2 ml) plus 3 ml of saline solution (Poliflex 0.9% isotonic 100 ml solution) plus 0,3 mg/kg of ketamine (Ketalar 500 mg). The impacted third molars of the patients will be removed.

The fourth group (Control group): Each patient in this group will be administered intravenous 100 ml saline (Poliflex 0.9% isotonic 100 ml solution) for a placebo effect 60 minutes before surgical third molar extraction. Before the procedure, patients will be given local anesthesia using a mixture of 2 ml of local anesthetic (Ultracain Ds Fort 2 ml) plus 3 ml of saline solution (Poliflex 0.9% isotonic 100 ml solution). The impacted third molars of the patients will be removed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a fully embedded third molar tooth in the mandible
* Patients with regular attendance for routine follow up
* Patients with a healthy general systemic condition

Exclusion Criteria:

* Patients with a fully erupted or partially embedded third molar tooth in the mandible
* Patients who have previously experienced allergies to NSAIDs, local anesthetics, and ketamine
* Pregnant or breastfeeding patients
* Patients who have recently used a different group of NSAIDs for a different condition

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
The pain level measurement after impacted third molar surgery will be assessed with the visual analog scale (VAS) in all groups. | The pain level measurements of all patients will be evaluated by a visual analog scale (VAS) two hours following impacted third molar surgery. [All study participants were asked to record their pain levels two hours after surgery].
  VAS (Pain intensity was assessed on a 100-mm visual analoge scale, where 0=no pain and 100=worst possible pain)
The pain level measurement after impacted third molar surgery will be assessed with the visual analog scale (VAS) in all groups. | The pain level measurements of all patients will be evaluated by a visual analog scale (VAS) six hours following impacted third molar surgery. [All study participants were asked to record their pain levels six hours after surgery].
  VAS (Pain intensity was assessed on a 100-mm visual analoge scale, where 0=no pain and 100=worst possible pain)
The pain level measurement after impacted third molar surgery will be assessed with the visual analog scale (VAS) in all groups. | The pain level measurements of all patients will be evaluated by a visual analog scale (VAS) 12 hours following impacted third molar surgery. [All study participants were asked to record their pain levels 12 hours after surgery].
  VAS (Pain intensity was assessed on a 100-mm visual analoge scale, where 0=no pain and 100=worst possible pain)
The pain level measurement after impacted third molar surgery will be assessed with the visual analog scale (VAS) in all groups. | The pain level measurements of all patients will be evaluated by a visual analog scale (VAS) 24 hours following impacted third molar surgery. [All study participants were asked to record their pain levels 24 hours after surgery].
  VAS (Pain intensity was assessed on a 100-mm visual analoge scale, where 0=no pain and 100=worst possible pain)
The limitation of mouth opening (trismus) after third molar surgery will be measured in all groups. | The limitation of mouth opening (trismus) after third molar surgery will be measured in all groups. [The maximum mouth opening of all study participants will be measured and recorded before surgery].
  Trismus was evaluated preoperatively by measuring the distance between the mesial-incisal corners of the upper and lower right central incisors at the maximum opening of the jaws.
The limitation of mouth opening (trismus) after third molar surgery will be measured in all groups | The limitation of mouth opening (trismus) after third molar surgery will be measured in all groups. [The maximum mouth opening of all study participants will be measured and recorded two days after the surgery].
  Trismus was evaluated on the second day postoperatively by measuring the distance between the mesial-incisal corners of the upper and lower right central incisors at the maximum opening of the jaws.
The limitation of mouth opening (trismus) after third molar surgery will be measured in all groups | The limitation of mouth opening (trismus) after third molar surgery will be measured in all groups. [The maximum mouth opening of all study participants will be measured and recorded seven days after the surgery].
  Trismus was evaluated on the seventh day postoperatively by measuring the distance between the mesial-incisal corners of the upper and lower right central incisors at the maximum opening of the jaws.

SECONDARY OUTCOMES:
The secondary outcome measure is the amount of rescue analgesia used by all participants after impacted third molar tooth surgery. | The mean amount of rescue analgesia used by all participants within the first 24 hours after surgery will be calculated.
  All study participants will record the dose of rescue analgesic medicine (Paracetamol 500 mg) at home if they need to take it within 24 hours following surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Faculty of Dentistry, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No